CLINICAL TRIAL: NCT02686242
Title: Influence of Spinal Anaesthesia on Hemodynamic Stability in Women With Placenta Previa Percreta Undergoing Caesarean Section
Brief Title: Spinal Aesthesia in Women With Placenta Previa Percreta
Acronym: SAW
Status: Completed | Type: Observational
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Zhihong LU, Dr., Air Force Military Medical University, China
Other Study IDs: XJH-A-2015-6-6-01
Record Dates: First submitted 2016-01-13; First posted 2016-02-19 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-06

CONDITIONS: Complications; Cesarean Section
Keywords: cesarean section; spinal anesthesia; general anesthesia
MeSH Terms: interventions — Anesthesia, Spinal; Anesthesia, General

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- spinal anesthesia: patients receive spinal anesthesia before general anesthesia
  Interventions: Procedure: spinal anesthesia
- general anesthesia: patients receive general anesthesia
  Interventions: Procedure: general anesthesia

INTERVENTIONS:
Procedure: spinal anesthesia — bupivacaine injected by spinal puncture
  Groups: spinal anesthesia
Procedure: general anesthesia — general anesthesia with intubation
  Groups: general anesthesia

SUMMARY:
Placenta previa percreta is a dangerous complication during surgery. Due to the high risk of hemorrhage, most parturients with placenta previa have to accept cesarean section. In this study investigators compare the effect of different anesthetic techniques on these patients.

ELIGIBILITY:
Inclusion Criteria:

* women with placenta previa and increta-percreta (diagnosed by ultrasound and/or magnetic resonance imaging and confirmed during cesarean section)
* women accepted cesarean section

Exclusion Criteria:

* women with baseline systemic blood pressure higher than 180 mmHg
* women with coagulation disorder

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: parturients with placenta praevia/accreta scheduled for cesarean section
Sampling Method: Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2015-12; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
incidence of hypotension | from beginning of the surgery to the end of the surgery,approximately 1 hour

SECONDARY OUTCOMES:
usage of norepinephrine | from beginning of the surgery to the end of the surgery,approximately 1 hour
dose of norepinephrine | from beginning of the surgery to the end of the surgery,approximately 1 hour
lowest systemic blood pressure | from beginning of the surgery to the end of the surgery,approximately 1 hour
maximal decrease of systemic blood pressure | from beginning of the surgery to the end of the surgery,approximately 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Hailong Dong, Study Chair — Xijing hosptial
Locations (1):
- Xijing Hospital, Fourth Military Medical University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kocaoglu N, Gunusen I, Karaman S, Ergenoglu AM, Firat V. Management of anesthesia for cesarean section in parturients with placenta previa with/without placenta accreta: a retrospective study. Ginekol Pol. 2012 Feb;83(2):99-103. PMID 22568353
- [Background] Ioscovich A, Mirochnitchenko E, Halpern S, Samueloff A, Grisaru-Granovsky S, Gozal Y, Einav S. Perioperative anaesthetic management of high-order repeat caesarean section: audit of practice in a university-affiliated medical centre. Int J Obstet Anesth. 2009 Oct;18(4):314-9. doi: 10.1016/j.ijoa.2009.01.014. Epub 2009 Aug 7. PMID 19665365
- [Background] Mok M, Heidemann B, Dundas K, Gillespie I, Clark V. Interventional radiology in women with suspected placenta accreta undergoing caesarean section. Int J Obstet Anesth. 2008 Jul;17(3):255-61. doi: 10.1016/j.ijoa.2007.11.010. Epub 2008 Jun 2. PMID 18513942